CLINICAL TRIAL: NCT01639521
Title: Randomized Phase II Trial Of Adjuvant Chemotherapy For Urothelial Carcinoma Comparing GC To Dose-Dense MVAC
Brief Title: Gemcitabine Hydrochloride and Cisplatin or High-Dose Methotrexate, Vinblastine, Doxorubicin Hydrochloride, and Cisplatin in Treating Patients With Urothelial Cancer
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Why Stopped: Lack of funding
Sponsor: University of Southern California (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 4B-10-5; NCI-2012-00961 (Registry Identifier: CTRP (Clinical Trial Reporting Program))
Record Dates: First submitted 2012-07-10; First posted 2012-07-12 (Estimated); Last update posted 2014-01-29 (Estimated); Status verified 2014-01

CONDITIONS: Anterior Urethral Cancer; Localized Transitional Cell Cancer of the Renal Pelvis and Ureter; Posterior Urethral Cancer; Recurrent Bladder Cancer; Recurrent Urethral Cancer; Regional Transitional Cell Cancer of the Renal Pelvis and Ureter; Stage III Bladder Cancer; Transitional Cell Carcinoma of the Bladder; Ureter Cancer; Urethral Cancer Associated With Invasive Bladder Cancer
MeSH Terms: conditions — Urinary Bladder Neoplasms; Urethral Neoplasms; Ureteral Neoplasms | interventions — Cisplatin; Gemcitabine; Methotrexate; merphos; Vinblastine; Doxorubicin; pegfilgrastim

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Arm A (gemcitabine hydrochloride, cisplatin) (Experimental): Patients receive cisplatin IV on day 1 and gemcitabine hydrochloride IV over 1 hour on days 1 and 8. Treatment repeats every 21 days for 4 courses in the absence of disease progression or unacceptable toxicity.
  Interventions: Drug: cisplatin; Drug: gemcitabine hydrochloride; Other: laboratory biomarker analysis
- Arm B (MVAC) (Experimental): Patients receive methotrexate IV on day 1 and vinblastine IV, doxorubicin hydrochloride IV, and cisplatin IV on day 2. Treatment repeats every 14 days for 4 courses in the absence of disease progression or unacceptable toxicity.
  Interventions: Drug: cisplatin; Drug: methotrexate; Drug: vinblastine; Drug: doxorubicin hydrochloride; Biological: pegfilgrastim; Other: laboratory biomarker analysis

INTERVENTIONS:
Drug: cisplatin — Given IV
  Other Names: CACP; CDDP; CPDD; DDP
Drug: gemcitabine hydrochloride — Given IV
  Other Names: dFdC; difluorodeoxycytidine hydrochloride; gemcitabine; Gemzar
  Arms: Arm A (gemcitabine hydrochloride, cisplatin)
Drug: methotrexate — Given IV
  Other Names: amethopterin; Folex; methylaminopterin; Mexate; MTX
  Arms: Arm B (MVAC)
Drug: vinblastine — Given IV
  Other Names: Velban; Velsar; VLB
  Arms: Arm B (MVAC)
Drug: doxorubicin hydrochloride — Given IV
  Other Names: ADM; ADR; Adria; Adriamycin PFS; Adriamycin RDF
  Arms: Arm B (MVAC)
Biological: pegfilgrastim — Given SC
  Other Names: Filgrastim SD-01; GCSF-SD01; Neulasta; SD-01 sustained duration G-CSF
  Arms: Arm B (MVAC)
Other: laboratory biomarker analysis — Correlative studies

SUMMARY:
This study is about two chemotherapy study drug combinations (regimens) that are used for urothelial (bladder or upper urinary tract) cancer. Both study drug regimens, gemcitabine (gemcitabine hydrochloride) plus cisplatin, and high-dose-intensity MVAC (methotrexate, vinblastine, doxorubicin plus cisplatin), are standard chemotherapy regimens. Both regimens are used to treat people with urothelial cancer that has spread to other organs. Both study drug regimens have been proven to be effective in lowering the risk of the cancer coming back, but it is not known which regimen is the best. This study hopes to learn whether there is a difference in the effectiveness and side effects of these two study drug regimens when they are given to people who have had their urothelial cancer completely removed.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES

To estimate the difference in the rate of unacceptable toxicity for dose-dense methotrexate, vinblastine, doxorubicin, and cisplatin (MVAC) and gemcitabine and cisplatin (GC) in the adjuvant treatment of urothelial cancer.

SECONDARY OBJECTIVES

To compare rates of disease recurrence at 3 years between dose-dense MVAC and GC.

To determine whether molecular markers excision repair cross-complementing-1 (ERCC-1) ribonucleoside-diphosphate reductase M-1 (RRM-1), breast cancer 1 (BRCA1) topoisomerase 2-alpha (Top2A) and protein 53 (p53) can predict those patients more likely to benefit from chemotherapy.

To investigate the potential utility of cytidine deaminase (CDA), ERCC-1, xeroderma pigmentosum group D (XPD), glutathione S-transferase P-1 (GSTP-1) and glutathione S-transferase M-1 (GSTM-1) as molecular markers which predict occurrence of significant toxicity during adjuvant chemotherapy for urothelial cancer.

OUTLINE: Patients are randomized to 1 of 2 treatment arms.

ARM A: Patients receive cisplatin intravenously (IV) on day 1 and gemcitabine hydrochloride IV over 1 hour on days 1 and 8. Treatment repeats every 21 days for 4 courses in the absence of disease progression or unacceptable toxicity.

ARM B: Patients receive methotrexate IV on day 1, vinblastine IV, doxorubicin hydrochloride IV, cisplatin IV on day 2 and pegfilgrastim subcutaneously (SC) on day 3. Treatment repeats every 14 days for 4 courses in the absence of disease progression or unacceptable toxicity. After completion of study treatment, patients are followed up every 3 months for 3 years.

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed high-grade urothelial carcinoma, stage T3bN0, T4N0 or any T stage with lymph node involvement, completely resected; including upper tract urothelial carcinoma
* The dominant histology must be transitional cell or urothelial but foci of other histologies less than 20 percent of the total tumor volume are permitted
* Absence of metastatic disease on radiographic imaging
* Patients must be enrolled and able to start treatment within 90 days of radical cystectomy or radical nephrectomy
* Creatinine less than institutional upper limit of normal (ULN) or clearance greater or equal to 50 mL/min (may be calculated by Cockcroft-Gault formula or measured from 24-hour urine collection)
* Serum total bilirubin less or equal to 1.5 x ULN (except for patients with Gilbert's)
* Alkaline phosphatase less or equal to 2.5 x ULN
* Serum glutamic oxaloacetic transaminase (SGOT) and serum glutamic pyruvate transaminase (SGPT) less or equal to 2.5 x ULN
* White blood cells (WBC) greater or equal to 3000
* Absolute neutrophil count (ANC) greater or equal to 1500
* Hemoglobin (Hb) greater or equal to 9
* Platelets greater or equal to 100,000
* Normal left ventricular ejection fraction, by echocardiogram or multi gated acquisition scan (MUGA)
* Patients must be recovered from surgery
* Eastern Cooperative Oncology Group (ECOG) performance status 0 or 1
* Willing and able to provide informed consent
* Willingness to use barrier contraception during study period

Exclusion Criteria:

* The presence of significant pleural effusion or ascites
* Prior systemic chemotherapy for urothelial carcinoma including neoadjuvant chemotherapy (prior intravesical therapy is permitted)
* History of malignancy within preceding 5 years, aside from non-melanoma skin cancer or previously treated or incidentally detected prostate cancer with undetectable PSA (after radical cystectomy or prostate cancer therapy)
* Peripheral neuropathy greater than grade 1
* The presence of active heart disease such as congestive heart failure or unstable angina

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2013-05; Primary Completion 2013-05 (Actual); Study Completion 2013-05 (Actual)

PRIMARY OUTCOMES:
Rate of unacceptable toxicity graded according to Common Terminology Criteria (CTC) v4.0 | Assessed up to 3 years
  80% confidence intervals (CI) will be constructed; for unacceptable toxicity, the confidence interval will be one-sided.

SECONDARY OUTCOMES:
Disease-free survival | From radical cystectomy to the time cancer recurrence is detected by clinical findings or during surveillance imaging, at 3 years

CONTACTS AND LOCATIONS:
Overall Officials: Tanya Dorff, Principal Investigator — University of Southern California